CLINICAL TRIAL: NCT05037331
Title: Improvement of the Value of Orally Administered Cancer Drugs: Arm 1: Osimertinib for Advanced EGFR-positive NSCLC Patients: A Phase II Study
Brief Title: Osimertinib for Advanced EGFR-positive NSCLC Patients
Status: Recruiting | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/00190
Record Dates: First submitted 2021-05-19; First posted 2021-09-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer; Non Small Cell Lung Cancer
Keywords: Osimertinib; advanced EGFR-positive; NSCLC; orally administered
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Lung cancer is the leading cause of cancer incidence (11.6%) and mortality (18.4%) globally[1]. Development of targeted therapies in the context of precision medicine changed the way lung cancer was diagnosed and treated. Small molecule inhibitors, like tyrosine kinase inhibitors (TKIs), are now standard first-line therapy for EGFR-positive non-small cell lung cancer (NSCLC). First-generation EGFR-TKIs gefitinib and erlotinib bind competitively to the ATP-binding site of EGFR TK domain. This binding in second-generation TKI afatinib is irreversible. These drugs have improved better outcome compared to standard conventional chemotherapy In spite of this, more than half of the patients with an EGFR TKI treatment develop resistance. Deletion in exon 19 and single point substitution L858R in exon 21 accounting for 44% and 41% of all EGFR mutations, respectively are the most common mutations in EGFR gene which cause this resistance in the patients. Asia has the highest prevalence of EGFR mutations (38.4%), followed by America (24.4%) and Europe (14.1%). Median progression-free survival of EGFR mutated NSCLC patients under erlotinib or gefitinib has been around 12 months and 5-year survival was 15%

DETAILED DESCRIPTION:
To evaluate the efficacy (Objective Response Rate), safety and tolerability of 80mg Osimertinib eod dosing in NSCLC patients with sensitizing EGFR mutations and/or EGFR T790M resistance mutation that have no prior EGFR treatment.

To investigate the efficacy and safety of Osimertinib 80mg/eod. Parameters like PFS, DoR, the incidence of brain metastases and OS will be assessed for the efficacy using RECIST criteria version 1.1. PFS in the brain will be another endpoint. Adverse events will be graded according to CTCAE v4.0 by recording vital signs, physical examinations, weight, ECG, ECOG performance status, clinical chemistry, haematology, urinalysis. We would use ctDNA to detect the mutations and compare the progress of the disease or the outcome of patients besides clinical assessments. The relationship between PK and selected efficacy, pharmacodynamic markers (like duration of inhibition of EGFR by hair follicle sampling) and safety endpoints will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study subjects should fulfil the following criteria:

  1. Provision of informed consent prior to any study-specific procedure
  2. Patients must be ≥ 18 years old
  3. Locally advanced /metastatic NSCLC not responsive to surgery or radiotherapy
  4. Validated activating EGFR sensitising mutations with or without T790M resistance mutation at the time of recruitment for patients who have no prior EGFR TKI treatment.
  5. Patients must be EGFR treatment naïve.
  6. ECOG Performance status is 0-1 with no deterioration over the last 2 weeks prior to study recruitment.
  7. Normal organ and bone marrow function measured within 28 days before the study as defined below:

     * Haemoglobin ≥ 9.0 g/dL and no blood transfusions in the 28 days prior to entry
     * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
     * No features suggestive of MDS/AML on peripheral blood smear
     * White blood cells (WBC) > 3x109/L
     * Platelet count ≥ 100 x 109/L
     * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
     * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
     * Serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN)
     * ECOG performance status 0-2
  8. A life expectancy ≥ 12 weeks in all patients.
  9. Females in childbearing age should be using adequate contraceptive measures, should not be breastfeeding and their pregnancy test prior to the start of treatment must be negative. Evidence of non-child-bearing potential is fulfilled by one of the following criteria at screening:

     * The post-menopausal period defined as age ≥50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
     * Women <50 years old they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range.
     * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not a tubal ligation
  10. Male patients should be willing to use barrier contraception
  11. The patient is willing to comply with the protocol during the study including undergoing treatment and scheduled visits and examinations including follow up.
  12. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and is considered suitable for accurate repeated measurements.

Exclusion Criteria:

* Patients should not enter the study if any of the following exclusion criteria are fulfilled:

  1. Treatment with other EGFR-TKI within 8 days or within five half-lives of the compound before study entry whichever is the longer; any cytotoxic chemotherapy, or other anticancer drugs against NSCLC within 14 days of study entry
  2. Previously treated with an immune checkpoint inhibitor
  3. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years
  4. Radiotherapy to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks before the study entry
  5. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of study treatment with the exception of alopecia grade 2 and platinum-related neuropathy.
  6. Unstable spinal cord compression/brain metastases unless asymptomatic and not requiring steroids for at least 2 weeks prior to the start of study treatment. For patients with brain metastases, gamma knife or stereotactic brain surgery is allowed prior to study treatment.
  7. Major surgery within 4 weeks of starting study treatment and patients must have recovered from any effects of any major surgery. Minor surgery is allowed.
  8. Patients currently receiving or unable to stop use medications or herbal supplements that are potent inhibitors of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 weeks prior). All patients must avoid concomitant use of any medications, herbal supplements and/or foods with known inducer/inhibitory effects on CYP3A4 unless part of protocol treatment.
  9. Severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which based on investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or having active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
  10. Past medical history of ILD, drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD
  11. Any of the following cardiac criteria:

      1. Mean resting corrected QT interval (QTc using Fredericia's formula) > 470 msec
      2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block)
      3. Any factors increasing the risk of QTc prolongation or arrhythmias such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
  12. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the drug or previous significant bowel resection that would preclude adequate absorption of Osimertinib
  13. History of hypersensitivity to Osimertinib (or drugs with a similar chemical structure or class to Osimertinib) or any excipients of these agents
  14. Males and females of reproductive potential who are not using an effective method of contraception and females who are pregnant or breastfeeding or have a positive serum pregnancy test prior to study entry
  15. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
  16. Previous allogeneic bone marrow transplant.

Ages: 21 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Osimertinib for Advanced EGFR-positive NSCLC Patients
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To investigate the safety of Osimertinib 80mg/eod using TCAE v4.0 | 4
  To investigate the safety of Osimertinib 80mg/eod using TCAE v4.0 To investigate the safety of Osimertinib 80mg/eod. Parameters like PFS, DoR, the incidence of brain metastases and OS will be assessed for the efficacy using RECIST criteria version 1.1. PFS in the brain will be another endpoint. Adverse events will be graded according to CTCAE v4.0 by recording vital signs, physical examinations, weight, ECG, ECOG performance status, clinical chemistry, haematology, urinalysis. We would use ctDNA to detect the mutations and compare the progress of the disease or the outcome of patients besides clinical assessments. The relationship between PK and selected efficacy, pharmacodynamic markers (like duration of inhibition of EGFR by hair follicle sampling) and safety endpoints will be assessed as well.

CONTACTS AND LOCATIONS:
Overall Officials: Goh, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore